CLINICAL TRIAL: NCT05524428
Title: Eliminating Barriers to Colorectal Cancer Screening Using Rapid Cycle Testing: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adjoa Anyane-Yeboa, M.D., Gastroenterologist // Instructor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 22167; P50CA244433 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Colo-rectal Cancer
Keywords: colorectal cancer; cancer; screening; implementation science; health equity; cancer equity; healthcare access; minority health; early detection; public health; health justice; rapid testing
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The investigators will use a mixed methods approach involving qualitative focus groups with health center providers and staff to identify barriers and facilitators to screening, and implementation science methods to test multilevel implementation strategies at the health centers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Introduction of Implementation Strategies (Other): The investigators will determine the best intervention and strategy (and thus implementers) based on high ranking barriers/facilitators identified in focus groups. A minimum of 2 implementation strategies will be developed and implemented at each level (patient, provider, system) at each site that considers (1) implementation strategy; (2) mechanism in which the strategy impacts the identified determinant (3) the determinant; (4) moderators that may influence the impact of the strategy; (5) the preconditions necessary for successful implementation; and (6) implementation outcomes affected. Each community health center (CHC) will serve as its own separate subject, and individual strategies will be tested using single case experimental design (SCED) at each CHC using component analysis to rapidly test and optimize our strategies. In SCED each subject serves as their own control, an intervention is systematically introduced and withdrawn, and the effects of the intervention are measured.
  Interventions: Behavioral: Implementation Science Strategy
- Withdrawal of Implementation Strategies (No Intervention): In SCED each subject serves as their own control, an intervention is systematically introduced and withdrawn, and the effects of the intervention are measured.

INTERVENTIONS:
Behavioral: Implementation Science Strategy — The investigators will be conducting focus groups and identifying barriers and facilitators, and the investigators will be matching identified barriers and facilitators to implementation strategies at the patient, provider, and system level which the investigators will be testing using rapid-cycle methods.
  Arms: Introduction of Implementation Strategies

SUMMARY:
The investigators will use a mixed methods study i.e. focus groups involving CHC staff as well as quantitative study which involves analyzing data that is available from the EHR and DRVS population management platform.

DETAILED DESCRIPTION:
Aim 1: Describe the demographics of the populations aged 45 - 49, 50-4, and over 55 to understand baseline screening needs and disparities.

Overview: The investigators will characterize the population in these age groups in order to understand resources needed to screen patients at age 50 and to expand screening to the USPSTF's draft guideline if passed.

Setting: The investigators will select 4 CHCs with distinctly diverse populations for Aim 1 and Aim 2.

Approach: The investigators will examine data from the EHR and the DRVS platform to determine: (1) the size and demographics of the three age groups; (2) the frequency in which this population presents to the CHC for primary care and other visits; and (3) current screening initiation patterns. Based on the findings of the investigator's initial evaluation, the investigators will estimate the additional colorectal cancer screening tests that will be required to screen this population promptly at age 50 and the additional resources that will be needed at each health center to meet this need. The investigators will also estimate the impact of a lower age of screening initiation. Analysis will be stratified by race/ethnicity, gender, age and insurance status to assess for any disparities that might be present.

Data Collection and Management: The DRVS population management platform provides the data needed to evaluate Aim 1. The Implementation Science Center for Cancer Control Equity (ISCCCE) data management team will pull the data needed for the participating CHCs, once selected. The investigators have existing data use agreements that will be amended for this specific project. Data flows and management procedures have already been established and will serve to expedite this study.

Aim 2: Conduct focus groups with key personnel to identify barriers and facilitators to screening in 4 different health centers with uniquely diverse populations.

Overview: The investigators will conduct focus groups to understand barriers and facilitators to colorectal cancer screening including perceptions around the change in screening age, attitudes about specific strategies to facilitate colorectal cancer screening (e.g. use of technological-based solutions to prompt screening, task shifting with integration of medical assistants into the screening process), proposed strategies to improve screening at the health center, and other likely barriers and facilitators.

Approach: The investigators will conduct focus groups with key personnel at the 4 participating health centers. The investigators will include an administrative leader and population health managers, data analysts and quality improvement staff, as well as nurse/practice managers, medical assistants, and providers (MD, NP, and/or PA). Focus groups will address: (1) barriers and facilitators to timely screening initiation; (2) perceptions around using technological solutions to prompt colorectal cancer screening; and (3) perceptions about task-shifting with integration of the medical assistants into the colorectal cancer screening process. Distinct barriers and facilitators/determinants will be identified at the patient, provider and system-level. These determinants will be prioritized (high, medium, low) based on number of times referenced in the interviews.

Data Analysis: Focus group data will be analyzed to identify key themes related to barriers and facilitators to screening.

Outcomes: The outcome of this aim will be identified barriers and facilitators to colorectal cancer screening at health centers with a key focus on understanding perceptions around utilization of technological solutions (e.g. pre-existing text message platforms at health centers, electronic registries) and integration of the medical assistants into the CRC screening workflow.

Aim 3: Develop and test intervention components to anticipate and address barriers and facilitators at the patient, provider and system-level using rapid cycle methods.

Overview: We will identify implementation strategies at patient, provider and systems-levels and match to identified Aim 2 barriers and facilitators, use design probes to understand the workflows and preconditions for implementation strategies, and individually test strategies using rapid cycle methods.

Approach:

* Development of Implementation Strategies: High ranking barriers from Aim 2 will be matched with implementation strategies that are most likely to influence implementation outcomes. A minimum of 2 implementation strategies will be developed at each level. When identifying strategies, we will consider the: (1) implementation strategy; (2) mechanism in which the strategy impacts the identified determinant (3) the determinant; (4) moderators that may influence the impact of the strategy; (5) the preconditions necessary for successful implementation; and (6) implementation outcomes affected.
* Design Probes: We will conduct design probes to understand the culture, climate and preconditions to implementation at each health center. We will use design probes to further understand the day-to-day workings at the health center and workflows. We will further tailor our implementation strategies based on additional barriers and facilitators that are identified from design probes.
* Rapid Cycle Testing: Individual strategies will be tested using single case experimental design (SCED). In SCED each subject serves as their own control, an intervention is systematically introduced and withdrawn, and the effects of the intervention are measured. For our study each CHC will serve as a separate subject. We will conduct a series of single case experiments at each CHC using component analysis to rapidly test and optimize our strategies. Component analysis allows researchers to assess several interventions or components of an intervention individually or as a treatment package in multiple assessments. A minimum of 2 strategies at each level (patient, provider, system) will be tested at each clinic site. For example, a patient-level strategy might include text messaging to patients, which is enabled by the DRVS platform. We might test whether single or multiple text messages around a patient's birthday can prompt screening uptake, or if messages prior to a health care visit increases uptake of screening offered. An example at the provider-level might include the impact of a motivational training if staff identify difficulty motivating patients as a barrier. A systems-level strategy might include incorporating CRC screening into the workflows of the health center using the medical assistants, if provider time limitations are identified as a barrier.
* Post-Implementation Survey: When implementation testing ends, our team will send out a survey to any CHC staff member (administrative leader and population health managers, data analysts and quality improvement staff, as well as nurse/practice manager, medical assistant, and provider [MD, NP, and/or PA]) involved with the implementation of strategies at the health center level, and the survey information we will collect will assess perceptions on feasibility, appropriateness, and acceptability of the implementation strategy used.

ELIGIBILITY:
Inclusion Criteria:

* Staff members at partnering sites (see locations) who are administrative leaders, population health managers, data analysts, quality improvement staff, nurses, nurse managers, practice managers, medical assistants, and providers.
* Staff members at partnering sites ages 18+.

Exclusion Criteria:

* Staff members that are not involved in CRC screening practices at CHCs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: Acceptability of Implementation Strategies | 4 months
  The investigators will measure the acceptability of the implementation strategies determined in Aim 2. This will be measured through a post-implementation survey given to the CHC staff members who participate in systems-level implementation at the two CHC pilot test sites in Aim 3.
Primary Outcome 2: Feasibility of Implementation Strategies | 4 months
  The investigators will measure the feasibility of the implementation strategies determined in Aim 2. This will be measured through a post-implementation survey given to the CHC staff members who participate in systems-level implementation at the two CHC pilot test sites in Aim 3.
Primary Outcome 3: Appropriateness of Implementation Strategies | 4 months
  The investigators will measure the appropriateness of the implementation strategies determined in Aim 2. This will be measured through a post-implementation survey given to the CHC staff members who participate in systems-level implementation at the two CHC pilot test sites in Aim 3.

SECONDARY OUTCOMES:
Secondary Outcome: CRC Screening Rates | 4 months
  The secondary outcomes will be change in colorectal cancer screening rate. This will be measured by the difference in the colorectal cancer screening tests ordered and completed compared to the pre-implementation period.

CONTACTS AND LOCATIONS:
Overall Officials: Adjoa Anyane-Yeboa, MD, MPH, Principal Investigator — Mass General Hospital // Harvard Medical School
Locations (4):
- United States (4):
  - Codman Square Health Center, Boston, Massachusetts
  - Brockton Neighborhood Health Center, Brockton, Massachusetts
  - East Boston Neighborhood Health Center, East Boston, Massachusetts
  - Duffy Health Center, Hyannis, Massachusetts

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.

REFERENCES:
- [Background] Roundtable NCC. Data & Progress. National Colorectal Cancer Roundtable; 2020.
- [Background] Siegel RL, Miller KD, Goding Sauer A, Fedewa SA, Butterly LF, Anderson JC, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2020. CA Cancer J Clin. 2020 May;70(3):145-164. doi: 10.3322/caac.21601. Epub 2020 Mar 5. PMID 32133645
- [Background] Siegel RL, Fedewa SA, Anderson WF, Miller KD, Ma J, Rosenberg PS, Jemal A. Colorectal Cancer Incidence Patterns in the United States, 1974-2013. J Natl Cancer Inst. 2017 Aug 1;109(8):djw322. doi: 10.1093/jnci/djw322. PMID 28376186
- [Background] Roundtable NC. American Cancer Society. Accessed November 5, 2020, https://nccrt.org/what-we-do/80-percentby-2018/
- [Background] Ahnen DJ, Wade SW, Jones WF, Sifri R, Mendoza Silveiras J, Greenamyer J, Guiffre S, Axilbund J, Spiegel A, You YN. The increasing incidence of young-onset colorectal cancer: a call to action. Mayo Clin Proc. 2014 Feb;89(2):216-24. doi: 10.1016/j.mayocp.2013.09.006. Epub 2014 Jan 4. PMID 24393412
- [Background] Wolf AMD, Fontham ETH, Church TR, Flowers CR, Guerra CE, LaMonte SJ, Etzioni R, McKenna MT, Oeffinger KC, Shih YT, Walter LC, Andrews KS, Brawley OW, Brooks D, Fedewa SA, Manassaram-Baptiste D, Siegel RL, Wender RC, Smith RA. Colorectal cancer screening for average-risk adults: 2018 guideline update from the American Cancer Society. CA Cancer J Clin. 2018 Jul;68(4):250-281. doi: 10.3322/caac.21457. Epub 2018 May 30. PMID 29846947
- [Background] Force USPST. Draft Recommendation Statement: Colorectal Cancer Screening. U.S. Preventive Services Task Force; 2020.
- [Background] Brown T, Lee JY, Park J, Nelson CA, McBurnie MA, Liss DT, Kaleba EO, Henley E, Harigopal P, Grant L, Crawford P, Carroll JE, Alperovitz-Bichell K, Baker DW. Colorectal cancer screening at community health centers: A survey of clinicians' attitudes, practices, and perceived barriers. Prev Med Rep. 2015 Sep 21;2:886-91. doi: 10.1016/j.pmedr.2015.09.003. eCollection 2015. PMID 26844165
- [Background] Lasser KE, Ayanian JZ, Fletcher RH, Good MJ. Barriers to colorectal cancer screening in community health centers: a qualitative study. BMC Fam Pract. 2008 Feb 27;9:15. doi: 10.1186/1471-2296-9-15. PMID 18304342
- [Background] O'Malley AS, Beaton E, Yabroff KR, Abramson R, Mandelblatt J. Patient and provider barriers to colorectal cancer screening in the primary care safety-net. Prev Med. 2004 Jul;39(1):56-63. doi: 10.1016/j.ypmed.2004.02.022. PMID 15207986
- [Background] Matthews BA, Anderson RC, Nattinger AB. Colorectal cancer screening behavior and health insurance status (United States). Cancer Causes Control. 2005 Aug;16(6):735-42. doi: 10.1007/s10552-005-1228-z. PMID 16049812
- [Background] Dallery J, Raiff BR. Optimizing behavioral health interventions with single-case designs: from development to dissemination. Transl Behav Med. 2014 Sep;4(3):290-303. doi: 10.1007/s13142-014-0258-z. PMID 25264468
- [Background] Ward-Horner J, Sturmey P. Component analyses using single-subject experimental designs: a review. J Appl Behav Anal. 2010 Winter;43(4):685-704. doi: 10.1901/jaba.2010.43-685. PMID 21541152